CLINICAL TRIAL: NCT02393274
Title: Investigation of Microcirculation in Patients With Venoarterial Extracorporeal Membrane Oxygenation Life Support
Brief Title: Microcirculation in Venoarterial Extracorporeal Membrane Oxygenation Life Support
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201412045RINA
Record Dates: First submitted 2015-03-15; First posted 2015-03-19 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2016-12

CONDITIONS: Heart Failure; Respiratory Failure
MeSH Terms: conditions — Heart Failure; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 28-day Survival: survive for at least 28 days after placement of extra-corporeal membrane oxygenation life support
  Interventions: Device: Extra-corporeal membrane oxygenation life support
- 28-day Nonsurvival: not survive for 28 days after placement of extra-corporeal membrane oxygenation life support
  Interventions: Device: Extra-corporeal membrane oxygenation life support

INTERVENTIONS:
Device: Extra-corporeal membrane oxygenation life support — venoarterial extra-corporeal membrane oxygenation life support

SUMMARY:
Extra-corporeal membrane oxygenation (ECMO) life support system can provide both cardiac and respiratory support to patients with heart and respiratory failure. It can save time for these organs to recovery or for these patients to receive further management. However, many patients will die in spite of ECMO support. One of the key factor is whether the blood flow provided by the ECMO can meet the requirement of organ perfusion. The adequacy of macrocirculation may be determined by arterial pressure and minute blood flow of ECMO. However, the adequacy of microcirculation remains as a major unresolved clinical problem. This is a prospective observational clinical trial. The sublingual microcirculation will be examined with the incident dark field video microscope within 6 hours after venoarterial ECMO placement, and then at 24 h, 48 h, 72 h, and 96 h. The severity of multiple organ injury and clinical data will be recorded as well. The major parameters of microcirculation include total small vessel density, perfused small vessel density, and microvascular flow index. The sublingual microcirculation will also be examined before weaning off ECMO, within 6 hours after ECMO removal, and then at 24 h, 48 h, and 72 h. Serum level of endothelial cell specific molecule-1 at specific time points will be examined. The data of 14-day mortality, 28-day mortality, duration of ECMO support, and intensive care unit stay will be recorded. This study aims primarily to investigate the relationship between microcirculation and prognosis of these patients. This study will also investigate the relationship among serum level of endothelial cell specific molecule-1, microcirculation, and prognosis of these patients. Wish the results of this study can be applied in further research to help to improve the quality of ECMO care.

ELIGIBILITY:
Inclusion Criteria:

* Patients who require venoarterial extra-corporeal membrane oxygenation (ECMO) life support

Exclusion Criteria:

* who can not take an examination of sublingual microcirculation within 6 hours after placement of venoarterial ECMO support
* Non-native speakers

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who require venoarterial extra-corporeal membrane oxygenation (ECMO) life support
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2015-04; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Perfused small vessel density | At enrollment (within 12 hour after placement of extra-corporeal membrane oxygenation life support)
  Perfused small vessel density measured by incident dark field video microscope

SECONDARY OUTCOMES:
Total small vessel density | At Enrollment
  Total small vessel density measured by incident dark field video microscope
Endocan level | At enrollment
Microvascular flow index | At enrollment
  Microvascular flow index measured by incident dark field video microscope

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chang Yeh, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Yeh YC, Lee CT, Wang CH, Tu YK, Lai CH, Wang YC, Chao A, Huang CH, Cheng YJ, Chen YS; NTUH Center of Microcirculation Medical Research (NCMMR). Investigation of microcirculation in patients with venoarterial extracorporeal membrane oxygenation life support. Crit Care. 2018 Aug 19;22(1):200. doi: 10.1186/s13054-018-2081-2. PMID 30121090